CLINICAL TRIAL: NCT00000629
Title: The Effects of Valproic Acid on Zidovudine Glucuronidation and Pharmacokinetics in HIV-Infected Patients.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 191
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2008-07-30 (Estimated); Status verified 2003-10

CONDITIONS: HIV Infections
Keywords: Valproic Acid; Zidovudine
MeSH Terms: conditions — HIV Infections | interventions — Valproic Acid; Zidovudine

INTERVENTIONS:
Drug: Valproic acid
Drug: Zidovudine

SUMMARY:
Primary objective: To study the pharmacokinetic interaction between zidovudine (AZT) and valproic acid in asymptomatic HIV-infected patients, characterizing AZT's oral bioavailability, plasma elimination half-time, plasma levels, and urinary excretion of AZT, 5'-O-glucuronide (GAZT), and 3'-amino-3'-deoxythymidine (AMT). Secondary objective: To establish the safety of short-term administration of AZT and valproic acid in combination with regard to hematologic parameters and liver function in asymptomatic HIV-infected patients.

Preliminary studies using human liver tissue have shown that valproic acid inhibits the metabolic inactivation of zidovudine (AZT), which may prolong the plasma half-life of AZT and thus prolong the duration of the drug's effects in the body.

DETAILED DESCRIPTION:
Preliminary studies using human liver tissue have shown that valproic acid inhibits the metabolic inactivation of zidovudine (AZT), which may prolong the plasma half-life of AZT and thus prolong the duration of the drug's effects in the body.

Six asymptomatic HIV-infected patients are treated with AZT orally every 8 hours on days 1 through 4, then with a single dose on day 5 (after 8 hours of fasting), followed by pharmacokinetic sampling. On days 6 through 9, patients receive AZT orally every 8 hours in combination with valproic acid (lowest dose in the first 5 patients and a higher dose in patients 6 and 7) orally every 8 hours. On day 10, AZT and 1 of the 2 doses of valproic acid are given orally as single doses, followed by pharmacokinetic sampling. AZT is continued alone orally every 8 hours on days 11 through 14, then resumed at the patient's usual dose beginning on day 15. Per 03/09/92 amendment, dosing schedule may be modified slightly to accommodate patients with scheduling conflicts.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

Vitamins if already being taken prior to start of therapy.

Patients must have:

* Asymptomatic HIV infection.
* CD4 count between 300 and 650.

Prior Medication:

Required:

* AZT at doses between 500 and 1200 mg/day for at least 6 weeks prior to enrollment.

Allowed:

* Aspirin, Tylenol, or ibuprofen up to 48 hours prior to start of therapy.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Positive Hepatitis B surface antigen or clinical evidence of chronic active hepatitis of any type.
* Signs or symptoms of HIV infection including oral candidiasis, history of multidermatomal zoster, unexplained weight loss in excess of 10 percent body weight in the past 6 months, chronic diarrhea, or history of AIDS-defining opportunistic infections.

Concurrent Medication:

Excluded:

* Concomitant medications (other than AZT) for the 14 days prior to start of therapy.

Patients with the following prior conditions are excluded:

* History of AZT intolerance including hematologic, hepatic, and/or neurologic toxicity.
* History of seizures.
* History of any antiepileptics within the past 10 years.
* History of abnormal bleeding or intrinsic or extrinsic coagulopathy.
* Signs or symptoms of HIV infection including oral candidiasis, history of multidermatomal zoster, unexplained weight loss in excess of 10 percent body weight in the past 6 months, chronic diarrhea, or history of AIDS-defining opportunistic infections.

Prior Medication:

Excluded:

* Antiepileptics within the past 10 years.
* Prior valproic acid.
* Concomitant medications (other than AZT) within 14 days of enrollment.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6

CONTACTS AND LOCATIONS:
Overall Officials: Lertora JJL, Study Chair
Locations (1):
- Tulane Univ Med School, New Orleans, Louisiana, United States

REFERENCES:
- [Background] Lertora J, Akula S, Greenspan D, Rege A, Agrawal K, George W, Hyslop N. Valproic acid inhibits zidovudine glucuronidation in patients with HIV infection. Int Conf AIDS. 1992 Jul 19-24;8(3):100 (abstract no PuB 7307)
- [Background] Lertora JJ, Rege AB, Greenspan DL, Akula S, George WJ, Hyslop NE Jr, Agrawal KC. Pharmacokinetic interaction between zidovudine and valproic acid in patients infected with human immunodeficiency virus. Clin Pharmacol Ther. 1994 Sep;56(3):272-8. doi: 10.1038/clpt.1994.137. PMID 7924122